CLINICAL TRIAL: NCT02741921
Title: Ability of Anesthesiologist to Placid a Double-lumen Tube. A Randomized Crossover Cadaver Study Comparing VivaSight DL and Conventional Double-lumen Tube
Brief Title: Conventional Double-lumen Tube vs VivaSight DL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 02/04/2016
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Endotracheal Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal airway (Experimental): intubation with normal airway Cormack-Lehane classivication I
  Interventions: Device: VivaSight DL; Device: conventional double-lumen tube
- difficult airway (Experimental): intubation with difficult airway Cormack-Lehane classivication III
  Interventions: Device: VivaSight DL; Device: conventional double-lumen tube

INTERVENTIONS:
Device: VivaSight DL — intubation using VivaSight DL tube
Device: conventional double-lumen tube — intubation using conventional double-lumen tube

SUMMARY:
The investigators sought to compare the time to intubation and success rate of the endotracheal intubation using standard double-lumen tube and video tube ETView DL in an adult cadaver model in normal and difficult airway conditions.

ELIGIBILITY:
Inclusion Criteria:

* fresh adult cadavers

Exclusion Criteria:

* cadavers with face injures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Time required for endotracheal intubation | 1 day
  time from pick up the tube to first ventilation

SECONDARY OUTCOMES:
Time required for visual confirmation of double lumen tube position position | 1 day
  Time required for visual confirmation of double lumen tube position position
success rate of intubation attempt | 1 day
  success rate of first intubation attempt
Ease of intubation | 1 day
  To access subjective opinion about the difficulty of each intubation method, participants were asked to rate it on a visual analog scale (VAS) with a score from 1 (extremely easy) to 10 (extremely difficult).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Department of Emergency Medicine, Warsaw, Masovia, Poland

REFERENCES:
- [Background] Kurowski A, Szarpak L, Truszewski Z, Czyzewski L. Can the ETView VivaSight SL Rival Conventional Intubation Using the Macintosh Laryngoscope During Adult Resuscitation by Novice Physicians?: A Randomized Crossover Manikin Study. Medicine (Baltimore). 2015 May;94(21):e850. doi: 10.1097/MD.0000000000000850. PMID 26020389
- [Background] Szarpak L, Kurowski A, Zasko P, Karczewska K, Czyzewski L, Bogdanski L, Adamczyk P, Truszewski Z. Double-lumen tube tracheal intubation in a manikin model using the VivaSight Double Lumen: a randomized controlled comparison with the Macintosh laryngoscope. Am J Emerg Med. 2016 Jan;34(1):103-4. doi: 10.1016/j.ajem.2015.10.018. Epub 2015 Oct 23. No abstract available. PMID 26527175